CLINICAL TRIAL: NCT06192173
Title: Comparison of Short- and Medium- Term Efficacy of Patent Foramen Ovale Closure and Medication in the Treatment of Migraine
Brief Title: Patent Foramen Ovale Closure in Migraine
Status: Completed | Type: Observational
Sponsor: Haiyan Wang (Other)
Responsible Party: Sponsor-Investigator, Haiyan Wang, Director, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022(078)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Migraine; Patent Foramen Ovale
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Closure group: Migraine patients with PFO who managed with percutaneous PFO closure.
  Interventions: Procedure: Percutaneous PFO closure
- Drug group: Migraine patients with PFO who treated with medicion.

INTERVENTIONS:
Procedure: Percutaneous PFO closure — Two kinds of interventional closure methods including DSA-guided and TEE-guided percutaneous intervention were performed on closure group.
  Groups: Closure group

SUMMARY:
The goal of this observational study is to retrospectively observe the effect of PFO closure and medication on migraine. The main questions it aims to answer are:

* Whether PFO closure is more effective in the treatment of migraine than traditional medical treatment
* What factors affect the effectiveness of migraine treatment ?

Participants will undergo contrast transthoracic echocardiography to diagnose PFO and evaluate right-to-left shunt. They will be treated with medication and PFO closure respectively according to guidelines. HIT-6 and a questionnaire about migraine were obtained at the baseline and repeated at the 6-month and 12-month follow-up visits.

Researchers will compare closure group and drug group to see efficacy of two groups in treating migraine.

DETAILED DESCRIPTION:
Migraine patients with PFO who were admitted to our hospital from January 2018 to August 2021 were enrolled.They will be treated with medication and PFO closure respectively according to guidelines. Headache impact test (HIT-6) and a questionnaire about migraine were obtained at the baseline and repeated at the 6th and 12th month follow-up visits.

1. HIT-6 was used to assess migraine severity.
2. Questionnaire included questions regarding average duration of migraine, migraine frequency, relief of migraine after treatment, family history and medication use.
3. △HIT-6 is the difference between baseline and follow-up in HIT-6 and is used to assess migraine relief. The days of migraine attacks per month (MAD) were calculated by the product of the frequency of headache attacks and average duration of each attack. Therefore, the days of migraine remission per month (MRD)= MAD at the 6th or 12th month follow-up- MAD at baseline. In comparison with baseline, 50% decrease in the number of total attacks was considered responder.
4. Four parameters were selected to evaluate the treatment effect: HIT-6, △HIT-6, MRD, and response rate.

ELIGIBILITY:
Inclusion Criteria:

Closure group:

* Migraine patients with grade II-III RLS of PFO confirmed by cTTE.
* HIT-6≥50.
* Meeting the surgical indications of PFO closure according to Chinese expert consensus on Prophylactic Closure of Patent foramen ovale published in March 2017
* Patients who have underwent PFO closure.

Drug group:

* Migraine patients with grade II-III RLS of PFO confirmed by cTTE.
* HIT-6 ≥ 50.
* Patients who have underwent drug treatment for 12 months.

Exclusion Criteria:

* Congenital heart diseases, cardiomyopathy, heart failure, valvular heart disease, arrhythmia, severe hypertension or other heart diseases.
* Patients with serious complications after closure.
* Patients who have other known triggers of migraine.
* Patients with incomplete follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Migraine patients who diagnosed with PFO and HIT-6 ≥50
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Headache impact test (HIT-6) | After recruiting, HIT-6 will be assessed and reported up to 12 weeks.
  HIT-6 is a self-report assessment tool that covers six dimensions (pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress) and widely used in headache impact surveys. Scores range from 36-78, < 49 indicating no effect, 50~55 some effect, 56~60 a relatively large effect, and > 60 severe effect. The higher HIT-6, the more severe the impact of headache on patients.
The days of migraine remission (MRD) | After recruiting, MRD will be assessed and reported up to 12 weeks.
  The days of migraine attacks per month (MAD) were calculated by the product of the frequency of headache attacks and average duration of each attack. Therefore, the days of migraine remission per month (MRD)= MAD at the 6th or 12th month follow-up- MAD at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, China

IPD SHARING:
Plan to Share IPD: No